CLINICAL TRIAL: NCT05861804
Title: Analgesic Efficacy of Rhomboid Intercostal Nerve Block for Minimal Invasive Heart Surgery: A Randomized Controlled Clinical Trial
Brief Title: Analgesic Efficacy of Rhomboid Intercostal Nerve Block for Minimal Invasive Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022.462.IRB1.182
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Minimal Invasive Heart Surgery; Rhomboid Intercostal Nerve Block
Keywords: rhomboid intercostal nerve block; minimal invasive heart surgery; cardiac anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Block group (Experimental): Participants who will be receiving a rhomboid intercostal nerve block
  Interventions: Procedure: Rhomboid Intercostal Nerve Block
- Control group (No Intervention): Participant who will not be receiving any intervention

INTERVENTIONS:
Procedure: Rhomboid Intercostal Nerve Block — Before the induction of general anesthesia, under aseptic conditions, rhomboid intercostal nerve block will be performed with a single dose of 20 ml of %0,25 bupivacaine with ultrasound guidance, by the senior anaesthesiologist.
  Arms: Block group

SUMMARY:
The goal of this clinical trial is to test the analgesic efficacy of rhomboid intercostal nerve block (RINB) in patients undergoing minimal invasive heart surgery (MIHS). The main questions it aims to answer are:

* How will the total perioperative opioid consumption of the patients receiving RINB change?
* How will RINB effect the patients' numeric rating scores for pain in the postoperative 24-hour period?
* How will RINB effect the postoperative extubation times?
* How will RINB effect the length of intensive care unit (ICU) stays on the postoperative period?
* How will RINB effect the incidence of opioid related side effects?

Participants will be divided in two groups:

* Block group will receive a RINB before the surgery.
* Control group will not receive any nerve block. Researchers will compare the results between the groups to see the postoperative effects concerning opioid consumption as well as the pain scores, respiratory parameters and ICU length of stay of the patients receiving RINB for minimal invasive heart surgery.

The hypothesis of this study is that participants receiving RINB for MIHS will have a less total opioid consumption 24 hours postoperatively.

DETAILED DESCRIPTION:
Rhomboid intercostal nerve block (RINB) was first defined by Elsharkawy et al in 2016 proposing to provide analgesia for both the anterior and posterior hemithorax. Minimal invasive heart surgeries require a surgical incision of the lateral thoracic wall. In order to ease the postoperative pain of patients undergoing MIHS, some regional anaesthesia techniques have been tried but there is no consensus on the best method. This study aims to assess the analgesic efficacy of RINB for MIHS. The hypothesis is that participants receiving RINB for MIHS will have a less total opioid consumption 24 hours postoperatively. Also, the postoperative pain scores, respiratory parameters and ICU length of stay of the participants will be recorded. Participants will be divided in two groups. The block-group will receive a RINB preoperatively in the operating room. The control-group will not receive any nerve block. The participants will be followed 24 hours postoperatively and their total opioid consumption, numeric rating scores for pain, postoperative extubation times, length of ICU stays, incidence of opioid related side effects will be recorded. Also the participants and the surgical teams perioperative pain related satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-80 undergoing minimal invasive heart surgery

Exclusion Criteria:

* Allergy to local anaesthetics
* Chronic opioid use history
* Patients with psychiatric disorders
* Patients who are not open to communication
* Patients with chronic organ failure
* Patients that do not give consent
* Patients that need emergency surgery within the first 24 hours of the initial surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours post-surgery
  all consumed opioids will be converted in morphine equivalents and then added to reach the total dosage

SECONDARY OUTCOMES:
Numeric rating scale scores for pain | 24 hours post-surgery
  the scale between 0: no pain and 10:highes pain answered by the participants
Extubation time after surgery | 24 hours post-surgery
  measured in hours
Length of intensive care unit stay | 1 week follow up after surgery
  measured in hours
Opioid related side effects | 24 hours post surgery
  Nausea, vomiting, pruritis, respiratory depression assessed by yes/no questions

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Darçın, MD, Study Director — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from 6 months after publication for 5 years
Access Criteria: no access criteria